CLINICAL TRIAL: NCT03504761
Title: Prospective, Multi-Center Study of the ClariCore Optical Biopsy System in Patients Undergoing Transrectal Ultrasound (TRUS)-Guided Prostate Biopsy for Real-Time Tissue Evaluation
Brief Title: ClariCore System Used in Transrectal Ultrasound Guided Prostate Biopsy for Real-Time Tissue Evaluation
Acronym: SCORE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Precision Biopsy, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CIP-1010-B
Record Dates: First submitted 2018-04-06; First posted 2018-04-20 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Cellular Diagnosis, Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- ClariCore System (Experimental): ClariCore System study designed to obtain prostate biopsies utilizing real-time tissue classification with the ClariCore Optical Biopsy System.
  Interventions: Device: ClariCore Optical Biopsy System

INTERVENTIONS:
Device: ClariCore Optical Biopsy System — Demonstrate the efficacy and safety of the ClariCore System in obtaining prostate biopsies utilizing real-time tissue classification.
  Other Names: ClariCore System

SUMMARY:
The purpose of this study is to demonstrate the effectiveness and safety of the ClariCore System in obtaining prostate biopsies with device feedback that provides real-time tissue classification.

DETAILED DESCRIPTION:
The purpose of this study is to collect information on prostate biopsies using the ClariCore System. The ClariCore System is designed to improve how the biopsies are being collected from the prostate by using light sensors (fiber optics) that can see changes in the prostate tissue. Researchers will study the information collected from the light sensors to study a method that has been developed to tell the difference between normal and suspicious (possibly cancerous) prostate tissue during the biopsy. This information will be given to the doctor in real-time. From this study, researchers hope to learn if this method can tell the difference between normal and suspicious prostate tissue, and if this can improve the evaluation of prostate tissue (biopsies).

ELIGIBILITY:
Inclusion Criteria:

* Males > 22 years old
* Patient scheduled for TRUS-guided prostate biopsy based on standard of care urologic requirements to assess for tissue malignancy (abnormal Digital Rectum Examination, Prostate Specific Antigen kinetics, age, ethnicity, family history, etc.)
* Enrolling physician must have expectation that prostate dimensions will meet minimum prostate volume and height requirements that will be evaluated at start of biopsy procedure (i.e., Prostate volume > 20cc and height at least 22mm)
* Patient signs an Institutional Review Board approved, Informed Consent form to participate in the study prior to any study mandated determinations or procedure

Exclusion Criteria:

* Any anatomical or co-morbidity contraindications to TRUS prostate biopsy
* Acute painful perianal disorder (i.e. rectal abscess)
* Symptomatic, acute prostatitis
* Surgical absence of a rectum or the presence of a rectal fistula
* Patient has systemic infection or evidence of any surgical site infection (superficial or organ space), including active urinary tract infection
* Previous prostate intervention [Transurethral Prostatectomy (TURP) (bipolar, monopolar, laser)], Transurethral Microwave Thermotherapy (TUMT), High-Intensity Focused Ultrasound (HIFU), Cryo, Rezum, Urolift], not including previous prostate biopsy
* Current use of blood thinning agents for medical comorbidity which prohibits the cessation of use as typically required per standard of care (SOC) or history of a bleeding disorder (e.g. coagulopathy)
* Prior pelvic irradiation
* Actively receiving therapy for the treatment of cancer (except for patients on 5-alpha reductase inhibitors, or non-melanoma skin cancers that are managed nonsystemically)
* Actively receiving intravesical therapy or within 6 months of treatment for bladder cancer
* Patient has compromised immune system
* Active inflammatory bowel disease within the last 6 months
* Any condition, or history of illness or surgery that, in the opinion of the Investigator, might confound the results of the study or pose additional risks to the patient (e.g. significant cardiovascular conditions or allergies)
* Patient is not likely to comply with the protocol or follow up evaluation
* Patient is participating in a clinical trial of another investigational drug or device that may impact participation in this clinical study
* Patient is unable to provide legal Informed Consent

Min Age: 22 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Estimated)
Dates: Start 2018-04-25 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Validation of the tissue classification algorithm | At time of procedure
  Correlate histopathology of tissue biopsy core samples with the tissue classification algorithm results obtained at the time of the procedure to validate the tissue classification algorithm.

SECONDARY OUTCOMES:
Sensitivity and Specificity | At time of procedure
  The sensitivity and specificity of the ClariCore System will be calculated and reported.
Cancer Detection Rate | At time of procedure
  The cancer detection per core rate in the Targeted Cores that have been classified as suspicious will be determined and reported.

OTHER OUTCOMES:
Identification of New or Clinically Significant Disease | At time of procedure, at time of 7 day follow up
  The number of instances where a new or more clinically significant disease (Gleason 7 or greater) is diagnosed during collection of the Targeted Cores compared to the SOC Cores
Adverse Event Incidence | Up to 7 days post-procedure
  The cumulative incidence of adverse events related to the device or the procedure.
Serious Adverse Event | Up to 7 days post-procedure
  The cumulative incidence of serious adverse events (SAEs) related to the device or the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Neal Shore, M.D., Principal Investigator — Carolina Urologic Research Center/Atlantic Urology Clinics
Locations (6):
- United States (6):
  - The Urology Center of Colorado, Denver, Colorado
  - Brady Urological Institute, Johns Hopkins Hospital, Baltimore, Maryland
  - NYU Langone Urology Associates, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology of San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No